CLINICAL TRIAL: NCT02327377
Title: Predicting Treatment Outcomes in Pediatric Functional Abdominal Pain
Brief Title: Web-based Management of Pediatric Functional Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Lynn Walker, Professor of Pediatrics; Division Director, Adolescent & Young Adult Health, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140559
Record Dates: First submitted 2014-12-10; First posted 2014-12-30 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Gastrointestinal Disorders, Functional
Keywords: Irritable bowel syndrome; Intervention studies; Visceral pain; Chronic pain; Abdominal pain; Dyspepsia; Nausea; Nociception; Parents; Coping behavior; Anxiety; Depression; Catastrophization; Reinforcement (psychology); Self efficacy; Health services overutilization; Questionnaires; Self report; Health surveys; Prospective studies; Adolescent health; Mental health services; Health services accessibility; Health diaries; National Institute of Child Health & Human Development (US.); Telemedicine; E-Health; Web-based intervention; Parenting education
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Visceral Pain; Chronic Pain; Abdominal Pain; Dyspepsia; Nausea; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online Cognitive Behavior Therapy (Experimental): Online cognitive behavior therapy for coping with pain
  Interventions: Behavioral: Online Cognitive Behavior Therapy
- Online Education (Active Comparator): Educational information about pain
  Interventions: Behavioral: Online Education

INTERVENTIONS:
Behavioral: Online Cognitive Behavior Therapy
  Arms: Online Cognitive Behavior Therapy
Behavioral: Online Education
  Arms: Online Education

SUMMARY:
Functional abdominal pain (FAP), a pediatric pain condition without significant organic pathology, is a precursor to chronic pain and high healthcare utilization in young adulthood. This project aims to identify child and family characteristics that predict differential responses to a Cognitive Behavior Therapy intervention administered online to patients with FAP and their parents. The goal is to acquire scientific knowledge to guide individualized treatment of patients with FAP.

DETAILED DESCRIPTION:
The goal of our research is to identify individual differences in pediatric functional abdominal pain (FAP) that predict differential health outcomes and can be used to develop tailored approaches to the evaluation and treatment of FAP. Effective treatment of FAP is a critical public health issue because it is among the most common pain problems during childhood and prospectively predicts risk for chronic pain, disability, and frequent health service utilization (HSU) in early adulthood. Although cognitive behavior therapy (CBT) delivered by highly trained professionals in face-to-face sessions has been found to reduce pain in some FAP patients, such intensive resources are not generally available to the large population of FAP patients. This study will evaluate an alternative, more efficient approach to treating pediatric FAP. The study builds on and integrates recent work by two leading investigators in pediatric pain. First, in a prospective natural history study of pediatric onset FAP patients followed into late adolescence/early adulthood, PI Walker and colleagues identified three distinct patient profiles (i.e., Low Pain Adaptive, High Pain Adaptive, High Pain Dysfunctional) comprised of pain severity, pain cognitions, and affect at the time of the initial FAP evaluation in childhood. These profiles predicted chronic pain and related health outcomes at follow-up (FU) nearly a decade later. Patients with the High Pain Dysfunctional profile at baseline had the poorest symptom outcomes and also exhibited pro-nociceptive central pain modulation in laboratory pain testing at FU. The heterogeneity of the FAP pain profile groups suggests that they may differ in treatment needs and in the extent to which they benefit significantly more from adjunctive behavioral treatment as compared to usual care alone. Second, Co-Investigator Palermo developed and tested a CBT intervention delivered online (Web-based Management of Adolescent Pain; Web-MAP) which is an efficient, easily disseminated treatment that significantly reduced pain and disability in youth with a variety of chronic pain diagnoses in comparison to youth randomized to a usual care, wait-list control group. This study merges these lines of research into an innovative study that will, for the first time: (Aim 1) evaluate the efficacy of WebMAP administered to FAP patients and their parents; (Aim 2) evaluate baseline moderators of treatment response, including our previously validated FAP pain profiles, pro-nociceptive central pain modulation, and parent characteristics (protectiveness, modeling pain behavior, catastrophizing about the child's pain); and (Aim 3) evaluate potential mediators of the effect of WebMAP on health outcomes. Pediatric patients (n = 300) ages 11-17 years will be randomized to either WebMAP or a Usual Care (UC) control group following their initial subspecialty FAP evaluation. Assessments will be at baseline, mid- and post-treatment, and at 6- and 12-months post baseline. Study results will produce knowledge that can be used to more efficiently target interventions to FAP patients according to their individual needs and thereby extend evidence-based care to more patients and ultimately reduce overall costs of care.

ELIGIBILITY:
Inclusion Criteria:

* Referred for medical evaluation of abdominal pain of more than 3 months duration
* No prior diagnosis of organic disease that explains the pain
* Access to a computer and the internet

Exclusion Criteria:

* Presence of major medical condition (e.g., diabetes)
* Does not speak English
* Has a disability that precludes participation
* Does not have a participating parent/guardian
* Found to have significant organic disease (e.g., ulcerative colitis) in the medical evaluation

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 344 (Actual)
Dates: Start 2014-04; Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline somatic symptoms | 2 months after baseline
  Change from baseline somatic symptoms as measured by the Children's Somatization Inventory
Change from baseline abdominal pain | long-term follow-up (6 and 12 months after baseline)
  Change from baseline abdominal pain as measured by Abdominal Pain Index

SECONDARY OUTCOMES:
Change from baseline activity limitations | 2 months after baseline
  Change from baseline activity limitations as measured by the Patient Reported Outcomes Measurement Information System Pain Interference Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Walker, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walker LS, Stone AL, Han GT, Garber J, Bruehl S, Smith CA, Anderson J, Palermo TM. Internet-delivered cognitive behavioral therapy for youth with functional abdominal pain: a randomized clinical trial testing differential efficacy by patient subgroup. Pain. 2021 Dec 1;162(12):2945-2955. doi: 10.1097/j.pain.0000000000002288. PMID 34793406

DOCUMENTS (1):
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT02327377/ICF_000.pdf